CLINICAL TRIAL: NCT06392217
Title: Real-world Study of Incadronate in Breast Cancer Patients With Metastatic Bone Disease: clinIcal Efficacy and Safety
Brief Title: clinIcal Efficacy and Safety of Incadronate in Breast Cancer With Bone Metastases
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Chief physician, Fudan University
Other Study IDs: RELIEF
Record Dates: First submitted 2024-03-27; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Bone Metastases
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a real-world study to explore the efficacy and safety of incadronate in the treatment of breast cancer patients with bone metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or above;
2. Can understand the purpose of clinical trials and the benefits and risks, voluntarily participate in and sign the informed consent
3. The physical status score of the Eastern Cooperative Oncology Group (ECOG) was ≤3;
4. Histologically or cytologically confirmed breast cancer;
5. Imaging or histocytology confirmed bone metastases;
6. There were indications of useing Incadronate and no contraindications in the use of Incadronate;
7. New York Heart Association（NYHA）cardiac function grade ≤II, No serious heart disease;
8. All women of childbearing age, fertile men or their spouses did not plan to have children or donate sperm throughout the trial period until 6 months after the last dose, or voluntarily took effective contraceptive measures.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients with acute and chronic infections, or with other serious diseases at the same time, were judged not suitable for this study;
3. Other malignant tumors within 5 years (except the following cases: cured skin basal cell carcinoma, cervical carcinoma in situ, thyroid papillary carcinoma; A second primary cancer that has been eradicated and has not recurred within five years; Investigators have identified the primary tumor source of the metastases);
4. Mental illness or mental disorder, poor compliance can not cooperate with and describe treatment response;
5. There are serious organic diseases or major organ failure, such as decompensated heart, lung, liver, kidney failure, which can not tolerate treatment;
6. Patients with bleeding tendency;
7. The researcher believes that the patient has other conditions that are not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients with bone metastases
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who had at least one Skeletal-related event（SRE） | 12 months
  The proportion of patients who had at least one SRE within 12 months after initial treatment with infadronate (including pathological fractures, spinal cord compression, radiotherapy or surgery for bone metastases);
the time to first SRE | 12 months
  The time from the first treatment with infadronate to the first observation of any SRE
Adverse events | 12 months
  Incidence and classification of various adverse events of infadronate

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center; Department of Oncology, Shanghai Medical College, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No